CLINICAL TRIAL: NCT00321061
Title: VRC 011: A Phase I Clinical Trial of Intramuscular, Subcutaneous and Intradermal Administration of an HIV-1 Multiclade DNA Vaccine, VRC-HIVDNA016-00-VP, and an HIV-1 Multiclade Adenoviral Vector Vaccine,VRC-HIVADV014-00-VP, in Uninfected Adult Volunteers
Brief Title: Phase I Study of Vaccination Schedule of Experimental HIV Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060149; 06-I-0149
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-12-02

CONDITIONS: HIV Infections
Keywords: HIV Negative; Healthy; Immunity; Preventive; Virus; Healthy Volunteer; HV
MeSH Terms: conditions — HIV Infections; Virus Diseases

INTERVENTIONS:
Drug: VRC-HIVDNA016-00, VRC-HIVADV014-00

SUMMARY:
This study will test whether a vaccination schedule of experimental HIV vaccines is safe and whether it causes side effects in healthy adult volunteers. It will also compare the effects of vaccine injected into the muscle (intramuscular), just under the skin (subcutaneous), or into the skin (intradermal) and will monitor the social impact of being in an HIV vaccine study.

Healthy volunteers 18-50 years old may be eligible for this 42-week study. Participants are screened for antibodies to adenovirus, a common virus that causes upper respiratory infections, such as the common cold. Half of the participants selected will be positive and half will be negative for antibodies to the virus.

The vaccines used in this study are known as VRC-HIVDNA016-00-VP (called the "DNA vaccine") and VRC-HIVADV014-00-VP (called the "rAd5 vaccine"). The DNA vaccine codes for four HIV proteins. The rAd5 vaccine is made using an adenovirus that has been modified to contain DNA that codes for three HIV proteins. These vaccines cannot cause HIV or adenoviral infections.

Participants are randomly assigned to one of six possible vaccination schedules that include "prime" and "booster" vaccines. The first vaccinations prime the immune system and the immune response is then boosted later. The groups differ in the type of vaccines given (DNA vaccine prime with rAd5 booster or rAd5 prime with rAd5 booster), in how the vaccine is administered (intramuscularly, subcutaneously or intradermally) and in the schedule of administration. All shots are given in the upper arm. Subjects fill out a diary card at home for 5 days after each vaccination, recording their temperature and any symptoms. The cards are turned in to the clinic at the first visit after all 5 days are completed. Subjects return for clinic visits about 3 days after each prime vaccination and either come in or call the clinic about 7 days after the injection. They call a study nurse 1 or 2 days after the booster vaccination.

Participants have 15-20 clinic visits during the course of the study, depending on their vaccination schedule. At each visit, they are checked for health changes or problems, asked how they are feeling and if they have taken any medications or other treatments, including over-the-counter medicines, herbal supplements, etc. Blood and urine samples are collected at some visits. Subjects are tested for HIV several times and asked questions about their sexual behavior and drug use. Throughout the stu...

DETAILED DESCRIPTION:
STUDY DESIGN:

The VRC DNA vaccine and VRC recombinant adenoviral vector (rAd5) vaccine have been previously shown to elicit immune responses to HIV-1-specific peptides when administered intramuscularly (IM) alone and in prime-boost schedules. This Phase I, randomized, open-label exploratory study will evaluate the safety and tolerability and the immune responses when IM, subcutaneous (SC) or intradermal (ID) routes of administration are used for the priming vaccinations in a prime-boost schedule. The randomization will ensure that subjects with negative and positive screening adenovirus type 5 antibody (Ad5Ab) titers will be equally represented in each prime-boost schedule evaluated in the study. Group 1 subjects will receive three DNA prime vaccinations followed by a rAd5 boost vaccination and Group 2 subjects will receive one rAd5 prime vaccination followed by a rAd5 boost vaccination. It is also of interest to explore whether vaccination by SC or ID route alters the functional qualities of the immune response. About half of the subjects who screen for HIV vaccine studies at the VRC Clinic have negative Ad5Ab titer and half have positive Ad5Ab titers.

The hypotheses are: 1) IM, SC and ID are all safe routes of administration for both the DNA and rAd5 vaccines; 2) all regimens will elicit immune responses to HIV-1-specific peptides; 3) intradermal administration will allow a lower dosage of the DNA vaccine to be used for eliciting an immune response; and 4) rAd5 booster administered after a rAd5 prime will boost the cellular and humoral immune response. The primary objectives relate to evaluation of the safety and tolerability of the DNA and rAd5 vaccines when administered by IM, SC and ID routes. Secondary objectives are related to evaluation of the immunogenicity of the vaccines when administered by SC and ID routes as compared to the IM route and the social impact of participating in an HIV-1 vaccine trial. Exploratory evaluations of the immunogenicity of the vaccination regimens are also planned.

PROTOCOL DESCRIPTION:

VRC-HIVDNA016-00-VP (DNA vaccine) is composed of 6 closed, circular DNA plasmids that encode HIV-1 Gag, Pol and Nef (from clade B) and Env glycoprotein from clade A, clade B, and clade C; each plasmid comprises 16.67 percent (by weight) of the vaccine. VRC-HIVADV014-00-VP (rAd5 vaccine) is composed of 4 recombinant non-replicating adenoviral vectors that encode for HIV-1 Gag/Pol polyproteins (from clade B) and Env glycoprotein from clade A, clade B, and clade C, which are combined in a 3:1:1:1 ratio, respectively.

SUBJECTS:

Sixty healthy adult volunteers, 18 to 50 years old, 30 subjects with negative Ad5Ab titers (less than 1:12) and 30 subjects with positive Ad5Ab titers (greater than or equal to 1:12).

STUDY PLAN:

Subjects with negative and positive Ad5Ab titers will be equally randomized to the six prime-boost schedules evaluated in the study as shown in the schema below. All injections will be administered by a needle and syringe device appropriate for the route of administration specified.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

1. 18 to 50 years old.
2. Available for clinical follow-up through Week 42 of the study.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Complete an Assessment of Understanding prior to enrollment and verbalize understanding of all questions answered incorrectly.
5. Able and willing to complete the informed consent process.
6. Willing to receive HIV test results and willing to abide by NIH guidelines for partner notification of positive HIV results.
7. Willing to donate blood for sample storage to be used for future research.
8. Willing to discuss HIV infection risks and amenable to risk reduction counseling.
9. In good general health without clinically significant medical history.
10. Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) less than 40 within the 28 days prior to enrollment.

    Laboratory Criteria within 28 days prior to enrollment:
11. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men.
12. White blood cells (WBC) = 3,300-12,000 cells/mm (3).
13. Differential either within institutional normal range or accompanied by site physician approval.
14. Total lymphocyte count greater than or equal to 800 cells/mm3.
15. Platelets equal 125,000 - 550,000/mm (3).
16. Alanine aminotransferase (ALT) less than or equal to 1.25 x upper limit of normal.
17. Serum creatinine less than or equal to upper limit of normal.
18. Normal urinalysis defined as negative glucose, negative or trace protein, and no clinically significant blood in the urine.
19. Negative Food and Drug Administration (FDA)-approved HIV blood test.
20. Negative hepatitis B surface antigen.
21. Negative anti-HCV (hepatitis C virus antibody) and negative HCV PCR.

    Female-Specific Criteria:
22. Negative beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.
23. A female participant must meet any of the following criteria:

    * No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

Or

- Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 42 of the study,

Or

* Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 42 of the study by one of the following methods:
* condoms, male or female, with or without a spermicide
* diaphragm or cervical cap with spermicide
* intrauterine device
* contraceptive pills or patch, Norplant, Depo-Provera or other FDA-approved contraceptive method
* male partner has previously undergone a vasectomy.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

Women:

1. Woman who is breast-feeding or planning to become pregnant during the 42 weeks of study participation.

   Volunteer has received any of the following substances:
2. HIV vaccine in a prior clinical trial.
3. Immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past 3 months (with the exception of corticosteroid nasal spray for allergic rhinitis; topical corticosteroids for an acute uncomplicated dermatitis, short-acting beta-agonists in controlled asthmatics; or a course of corticosteroids that was 10 days or fewer in duration that was completed at least 2 weeks prior to study enrollment for a non-chronic condition).
4. Blood products within 120 days prior to HIV screening.
5. Immunoglobulin within 60 days prior to HIV screening.
6. Investigational research agents within 30 days prior to initial study vaccine administration.
7. Live attenuated vaccines within 30 days prior to initial study vaccine administration.
8. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration.
9. Current anti-tuberculosis prophylaxis or therapy.

   Volunteer has a history of any of the following clinically significant conditions:
10. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain.
11. Autoimmune disease or immunodeficiency
12. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.
13. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
14. History of thyroidectomy or thyroid disease that required medication within the past 12 months.
15. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years.
16. Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.
17. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
18. Syphilis infection that is active or a positive serology due to a syphilis infection treated less than six months ago.
19. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
20. Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.
21. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
22. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within five years prior to enrollment, history of a suicide plan or attempt.
23. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.
24. A subject with 3 or more of the 5 health risk factors noted below will be excluded:

    * Current smoker (or quit smoking less than 28 days prior to enrollment)
    * BMI greater than 35
    * Fasting low density lipoprotein (LDL) greater than 159 mg/dL or fasting cholesterol greater than 239 mg/dL
    * Systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
    * Fasting blood glucose greater than 125 mg/dL

Note: The fasting blood tests require 8 hours fast prior to the blood draw. The results used for eligibility screening must be from tests completed no more than 12 weeks (84 days) prior to day of enrollment. The individual criteria for BMI (inclusion item 10) and blood pressure (exclusion item 16) must also be met.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-04-25; Primary Completion 2009-12-02 (Actual); Study Completion 2009-12-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Osmanov S, Pattou C, Walker N, Schwardlander B, Esparza J; WHO-UNAIDS Network for HIV Isolation and Characterization. Estimated global distribution and regional spread of HIV-1 genetic subtypes in the year 2000. J Acquir Immune Defic Syndr. 2002 Feb 1;29(2):184-90. doi: 10.1097/00042560-200202010-00013. PMID 11832690
- [Background] Sugaya M, Lore K, Koup RA, Douek DC, Blauvelt A. HIV-infected Langerhans cells preferentially transmit virus to proliferating autologous CD4+ memory T cells located within Langerhans cell-T cell clusters. J Immunol. 2004 Feb 15;172(4):2219-24. doi: 10.4049/jimmunol.172.4.2219. PMID 14764689
- [Background] Peachman KK, Rao M, Alving CR. Immunization with DNA through the skin. Methods. 2003 Nov;31(3):232-42. doi: 10.1016/s1046-2023(03)00137-3. PMID 14511956
- [Derived] Enama ME, Ledgerwood JE, Novik L, Nason MC, Gordon IJ, Holman L, Bailer RT, Roederer M, Koup RA, Mascola JR, Nabel GJ, Graham BS; VRC 011 Study Team. Phase I randomized clinical trial of VRC DNA and rAd5 HIV-1 vaccine delivery by intramuscular (i.m.), subcutaneous (s.c.) and intradermal (i.d.) administration (VRC 011). PLoS One. 2014 Mar 12;9(3):e91366. doi: 10.1371/journal.pone.0091366. eCollection 2014. PMID 24621858